CLINICAL TRIAL: NCT06587737
Title: A Double-blind, Randomized, Placebo-controlled, Phase III Study for Reducing Dependency and Cardiovascular Events with Oral Colchicine 0.5mg Once Daily Compared with Placebo in Participants with Spontaneous Intracerebral Hemorrhage and Established, or Risk Factors For, Atherosclerosis
Brief Title: Colchicine for the Reduction of Dependency and Vascular Events After an Acute Intracerebral Hemorrhage
Acronym: CoVasc-ICH 2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CoVasc-ICH 2
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Colchicine; ICH - Intracerebral Hemorrhage; Stroke; Dependence
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, phase III study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- colchicine 0.5mg OD (Experimental)
  Interventions: Drug: Colchicine 0.5 MG
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — colchicine 0.5mg once-daily
  Arms: colchicine 0.5mg OD
Drug: Placebo — matching placebo, lacking active ingredient, once-daily
  Arms: placebo

SUMMARY:
Data indicate that patients with intracerebral hemorrhage (ICH) are at high risk for thromboembolic events and disability that is not being sufficiently mitigated by current treatment strategies. This is aggravated by the cessation of antithrombotic medications for significant periods after hemorrhage. These findings highlight the need for novel treatments that modify the high risk for major vascular events and functional outcomes in ICH survivors.

The objective of CoVasc-ICH 2 is to demonstrate that oral colchicine 0.5 mg daily is superior to placebo for improving the outcomes of ICH survivors with evidence or risk factors for atherosclerosis, when started within 72 hours from ICH onset.

ELIGIBILITY:
Inclusion Criteria:

Adult patients presenting with spontaneous intraparenchymal hemorrhage within 72 hours of symptom onset and qualifying for at least one of the following categories:

i. history of symptomatic coronary, peripheral and/or carotid artery disease (severe atherosclerotic vascular disease), or ii. visualized extracranial cervical/intracranial atherosclerotic disease causing any degree of stenosis/occlusion or presence of aortic arch plaque with maximum thickness ≥1 mm (moderate atherosclerotic vascular disease), or iii. two or more risk factors including: age 60 years or older, hypertension, dyslipidemia, diabetes mellitus, chronic kidney disease (eGFR: 15-50mL/min), history of ischemic stroke or current smoking (mild atherosclerotic vascular disease).

Exclusion Criteria:

* secondary causes of ICH (such as trauma, macrovascular anomalies, neoplasms or bleeding diathesis)
* ICH volume more than 60ml in the last imaging scan prior to consent
* Glasgow Coma Scale (GCS) score less than 7 or being intubated at the time of consent
* inflammatory bowel disease or chronic diarrhea
* cirrhosis or severe hepatic dysfunction
* renal insufficiency (eGFR<15mL/min)
* concurrent or planned treatment with strong CYP3A4 inhibitors (atazanavir, clarithromycin, darunavir/ritonavir, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, tipranavir/ritonavir) or P-gp inhibitors (cyclosporine, ranolazine)
* pregnancy or breast-feeding
* known allergy or sensitivity to colchicine
* a strong indication for colchicine where assignment to placebo is deemed unacceptable
* estimated life expectancy less than 6 months at the time of enrollment, and
* inability to adhere to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1125 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: MACE and Dependency | through study completion, an average of 36 months
  Treatment with colchicine will reduce the risk for major adverse cardiovascular events (MACE) and dependency
Safety: Symptomatic hematoma expansion, major gastrointestinal adverse reactions or infection rates | through study completion, an average of 36 months
  There will be no clinically-important change in symptomatic hematoma expansion, major gastrointestinal adverse reactions or infection rates with oral colchicine 0.5mg OD compared with matching placebo

CONTACTS AND LOCATIONS:
Overall Officials: Aristeidis Katsanos, MD, Principal Investigator — Population Health Research Institute, Hamilton Health Sciences, McMaster University; Ashkan Shoamanesh, MD, Principal Investigator — Population Health Research Institute, Hamilton Health Sciences, McMaster University

IPD SHARING:
Plan to Share IPD: Undecided